CLINICAL TRIAL: NCT03961828
Title: Evaluation of Liver Fibrosis by Serum Hyalornic Acid Measurement in β-Thalassemic Children Infected With Hepatitis C Virus Before and After Direct-Acting Antiviral Therapy
Brief Title: Hyalornic Acid Level in β-Thalassemic Children Treated for Hepatitis C Virus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eslam Elhawary, Lecturer of pediatric hemato-oncology and bone marrow transplantation, Tanta University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31747/08/17
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Beta-Thalassemia; Hepatitis C
MeSH Terms: conditions — beta-Thalassemia; Hepatitis C | interventions — ledipasvir; Sofosbuvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thalassemia with HCV (Experimental): The study was carried out upon 50 β-thalassaemic children infected with hepatitis C virus who attended for a medical check-up at the Hematology Unit, Pediatric Department, Tanta University Hospital. Hepatitis C virus infection was diagnosed by serological detection of HCV-Ab, and quantitative detection of serum HCV RNA by polymerase chain reaction (PCR).
  Interventions: Drug: Ledipasvir 90 MG / Sofosbuvir 400 MG [Harvoni]

INTERVENTIONS:
Drug: Ledipasvir 90 MG / Sofosbuvir 400 MG [Harvoni] — The fifty (50) thalassemic children infected with HCV received the new direct-acting antiviral therapy in the form of Ledipasvir (90 mg)/Sofosbuvir (400 mg); (Harvoni) as a single oral tablet /day for 12 weeks Follow up of these patients was performed for 24 weeks. Re-evaluation of these children after 24 weeks from initiation of Ledipasvir/Sofosbuvir treatment was performed by repeating clinical assessment, Fibroscan of liver , laboratory investigations including quantitative HCV RNA by PCR and serum hyaluronic acid measurement.
  Other Names: Measuring level of Hyalornic Acid; Fibroscan of liver

SUMMARY:
Patients with transfusion dependent Beta Thalassemia suffer from a high incidence of Hepatitis C infection especially in developed countries as Egypt. In our patients we also found a high correlation between hepatitic C infection and Liver fibrosis. in this study we offer our patients treatment with Direct antiviral drugs and assessed the degree of fibrosis before and after treatment. We tested Hyalornic acid as a predictor of the degree of fibrosis before and after treatment.

DETAILED DESCRIPTION:
The thalassemias are a heterogeneous group of genetic heritable disorders of hemoglobin (Hb) synthesis, considered as the most common monogenic disorder in the world, affecting men and women equally and poses a severe health and economic burden to patients and families at risk (Mohammad and Al-Doski, 2012). Thalassemia is a major health problem in Egypt since it estimated out of 1.5 million live births, 1000 children with thalassemia are born annually (Youssef et al., 2012).

Thalassemics can develop liver fibrosis because of iron liver overload and hepatitis virus C (HCV) infection. Multicenter cross-sectional studies have reported that the development and the severity of liver fibrosis are strongly related to the extent of liver iron overload and to the presence of chronic HCV infection (Di Marco et al., 2008). HCV infection is the main risk factor for liver fibrosis in transfusion-dependent thalassemics. Excess liver iron is now clearly recognized as a cofactor for the development of advanced fibrosis in patients with HCV infection (Elalfy et al., 2013). Although, hepatic fibrogenesis has long been thought to be an irreversible process, it is now evident that it is a dynamic process with significant potential for reversal; unlike cirrhosis, which is irreversible. Identification of liver fibrosis at an early stage would be of great significance (Manning DS and Afdhal NH, 2008, Xu et al., 2003) Liver biopsy is an essential method for assessing fibrosis and it continues to have an important role in the diagnosis, prognosis, and management of patients with elevated results of iron studies and abnormal liver function test results. Therefore, liver biopsy is currently considered the gold standard for assessing hepatic fibrosis (Di Marco et al., 2008). However, it is an invasive and painful procedure, with rare but potential life threatening complications, limiting its acceptance and repetition in usually asymptomatic patients. In addition, the accuracy of liver biopsy in assessing fibrosis may be questioned because of sampling error and interobserver variability, which may lead to under or overstaging of fibrosis or cirrhosis (Foucher et al., 2006).

Thus there is a need to develop and validate non-invasive tests that can accurately reflect the full spectrum of hepatic fibrosis, cirrhosis, and its severity in liver diseases (Foucher et al., 2006). Serum markers and imaging methods are increasingly in vogue non-invasive alternatives to liver biopsy and the development of safe, inexpensive, and reliable non-invasive fibrosis measurement tools remains a research priority in clinical hepatology (Rockey DC 2006).

Hyaluronic acid (HA) is a high molecular weight glycosaminoglycan which is an essential component of extracellular matrix in almost every tissue in the body (Papastamataki, 2010). In the liver, HA is mostly synthesized by the hepatic stellate cells and removed via sinusoidal cell adhesion molecules (Halfon, 2005). This mechanism is impeded in fibrosis, leading to a rise in serum levels of HA. Therefore, serum HA is considered a marker that appears early before pathological changes occur (Zheng, 2003). Serum HA levels have been shown to correlate with histological stages of liver fibrosis in hepatitis C virus patients. Therefore, HA has a good diagnostic accuracy as a noninvasive assessment of fibrosis and cirrhosis (Parise et al, 2006).

Children with chronic hepatitis C (CHC) in are at risk for major complications, including cirrhosis, hepatocellular carcinoma, and death. The combined pegylated interferon-α and ribavirin (PEG-IFN/ribavirin) remains the standard therapy for CHC in children until 2016 (Aziz S, 2014, Suzuki et al. 2016, Yang et al 2017). The approved PEG-IFN/ribavirin therapy for children aged 3 and older is often held from use until adulthood because of its extensive list of potential side effects and high likelihood of causing adverse symptoms. In children and adolescents with HCV, treatment and reduction of the spread of HCV before adulthood is important, as there can be transmission to other individuals via sexual activity and infected females can later vertically transmit the infection during pregnancy, the latter representing a common source of transmission for children (Yang et al 2017).

In recent years, a number of direct-acting antiviral agents (DAAs) are under development for treatment of CHC. DAAs reduce the amount of HCV in the body by blocking viral replication inhibiting directly one of the several steps of HCV lifecycle preventing the virus from multiplying, and in most cases, they cure HCV. DAAs are classified into several categories based on their molecular target (Perales et al., 2015, Manns et al., 2016). The recent development of DAAs has shown promising results in clinical trials for use in children and adults and has dramatically increased the rates of sustained virological response (SVR) while improving side effect profiles as compared to interferon based treatments (Yang et al 2017). New DAAs available for adults have still not been approved for treatment in children (Aziz S, 2014, Serranti et al., 2014, Ohmer et al., 2016, Yang et al 2017). However, the approval of ledipasvir/sofosbuvir and sofosbuvir with ribavirin for adolescents is potentially anticipated as early as 2017 (Yang et al 2017).

Recently (on April 7, 2017), the U.S. Food and Drug Administration (FDA) approved the first DAAs for children that included sofosbuvir (Sovaldi) and sofosbuvir/ledipasvir (Harvoni) to treat HCV in children and adolescents aged 12 years and older or weighing at least 35 kilograms. These DAAs (Harvoni and Sovaldi) were previously approved to treat HCV in adults. These approvals will help change the landscape for HCV treatment by addressing an unmet need in children and adolescents (FDA News Release 2017, HCV Guidance 2017). The adult fixed-dose of ledipasvir/sofosbuvir resulted in similar plasma exposure of ledipasvir, sofosbuvir, and GS-331007 (the inactive metabolite of sofosbuvir) in adolescents as in adults, thus the adult dose was used for this age group (Schwarz et al. 2016). Similarly, giving half the adult fixed-dose of ledipasvir/ sofosbuvir, 45 mg/200 mg, to children ages 6-11 resulted in comparable plasma exposure of ledipasvir, sofobuvir, and GS-331007 as in adults, without any severe adverse events or laboratory abnormalities (Garrison et al 2016).

ELIGIBILITY:
Inclusion Criteria:

* β-thalassemic children with superadded hepatitis C virus infection

Exclusion Criteria:

1. Liver decompansatoin.
2. Children <12years old.
3. Patients with viral hepatitis B

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Treatment of Hepatitis C | 24 weeks
  Becoming PCR negative for Hepatitis C

SECONDARY OUTCOMES:
Reduction of liver fibrosis | 6 months
  improvement of Fibroscan and Hyalornic Acid Level significantly after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Hematology Unit, Faculty of Medicine, Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No